CLINICAL TRIAL: NCT06389786
Title: MC230504 Safe Omission of Pelvic Lymph Node Dissection (SOuND ) During Radical Prostatectomy: Diagnostic Accuracy of rhPSMA-7.3(18F) PET/CT, mpMRI and Patient Clinical Factors to Predict Lymph Node Metastasis
Brief Title: Accuracy of 18F-rhPSMA-7.3 PET/ MRI for Prediction of Lymph Node Metastasis in Localized High-Risk Prostate Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: MC230504; NCI-2024-03306 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 23-009377 (Other: Mayo Clinic Institutional Review Board); MC230504 (Other: Mayo Clinic)
Record Dates: First submitted 2024-04-25; First posted 2024-04-29 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Localized Prostate Carcinoma; Oligometastatic Prostate Carcinoma; Stage I Prostate Cancer AJCC v8; Stage II Prostate Cancer AJCC v8; Stage III Prostate Cancer AJCC v8; Stage IVA Prostate Cancer AJCC v8
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Specimen Handling; Robotics; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Screening (18F-rhPSMA-7.3 PET/MRI) (Experimental): Patients receive 18F-rhPSMA-7.3 IV and undergo PET/MRI up to 30 days prior to SOC robotic radical prostatectomy with bilateral pelvic lymph node dissection. Patients also undergo CT/MRI or bone scan/PT, as well as tissue collection during screening.
  Interventions: Procedure: Bilateral Pelvic Lymph Node Dissection; Procedure: Biospecimen Collection; Procedure: Bone Scan; Procedure: Computed Tomography; Other: Electronic Health Record Review; Other: Flotufolastat F-18 Gallium; Procedure: Laparoscopic Radical Prostatectomy with Robotics; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography

INTERVENTIONS:
Procedure: Bilateral Pelvic Lymph Node Dissection — Undergo bilateral pelvic lymph node dissection
Procedure: Biospecimen Collection — Undergo tissue sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Scan — Undergo bone scan
  Other Names: Bone Scintigraphy
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Other: Electronic Health Record Review — Ancillary studies
Other: Flotufolastat F-18 Gallium — Given IV
  Other Names: (18F)-rhPSMA-7.3; 18F-rhPSMA-7.3; 18FrhPSMA-7.3; F-18-rhPSMA-7.3; Fluorine F 18 Radiohybrid PSMA-7.3; Fluorine F 18 rhPSMA-7.3; Fluorine-18 rhPSMA-7.3; Posluma; rhPSMA-7.3 (18F)
Procedure: Laparoscopic Radical Prostatectomy with Robotics — Undergo robotic radical prostatectomy
  Other Names: RARP; Robot-assisted Radical Prostatectomy
Procedure: Magnetic Resonance Imaging — Undergo MRI or PET/MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Procedure: Positron Emission Tomography — Undergo PET/MRI
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT

SUMMARY:
This clinical trial evaluates the use of an imaging scan (18F-rhPSMA-7.3 positron emission tomography [PET]/magnetic resonance imaging [MRI]) for identifying patients who are at risk of having their disease spread to the lymph nodes in those undergoing radical prostatectomy for prostate cancer that has not spread to other parts of the body (localized). Prostate specific membrane antigen (PSMA) PET/computed tomography (CT) has emerged as an option to stage newly diagnosed high risk prostate cancer patients. PSMA PET/CT has demonstrated improved diagnostic accuracy for identifying metastasis. PET is procedure in which a small amount of radioactive glucose (sugar) is injected into a vein, and a scanner is used to make detailed, computerized pictures of areas inside the body where the glucose is used. Because cancer cells often use more glucose than normal cells, the pictures can be used to find cancer cells in the body. MRI is procedure in which radio waves and a powerful magnet linked to a computer are used to create detailed pictures of areas inside the body. These pictures can show the difference between normal and diseased tissue. This study may help researchers learn whether 18F-rhPSMA-7.3 PET/ MRI may improve predicting which patients are at risk of lymph node metastases and who are suitable candidates for pelvic lymph node dissection in patients with localized high-risk prostate cancer undergoing radical prostatectomy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To investigate the diagnostic ability of flotufolastat F-18 gallium (18F-rhPSMA-7.3) PSMA PET/MRI prior to radical prostatectomy in newly diagnosed, high-risk prostate cancer patients.

SECONDARY OBJECTIVES:

I. Calculating the specificity, positive-predictive value, and negative-predictive value for the detection of lymph node positivity.

II. Investigating the rates of biochemical recurrence (BCR) as measured by post-operative prostate specific antigen (PSA) (PSA > 0.20) at pre-defined timepoints in patients.

OUTLINE:

Patients receive 18F-rhPSMA-7.3 intravenously (IV) and undergo PET/MRI up to 30 days prior to standard of care (SOC) robotic radical prostatectomy with bilateral pelvic lymph node dissection. Patients also undergo CT/MRI or bone scan/PET, as well as tissue collection during screening.

Upon completion of study treatment, patients are followed up at 6 weeks, 3 months, 9 months, and 12 months post-surgery.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects ≥ 30 and ≤ 85 years old
* Primary diagnosis of prostate cancer selected for surgical intervention (radical prostatectomy with extended lymph node dissection)
* Primary diagnosis of untreated American Urological Association (AUA) guidelines high-risk localized prostate cancer, hormone-naïve prostate cancer via contrast enhanced prostate MRI + tissue sampling
* Planned elective radical prostatectomy with extended pelvic lymph node dissection
* Clinical oligometastatic disease with ≤ 3 nodes positive on preoperative standard of care imaging of prostate region within 6 months of surgery
* Patient agrees to comply with the investigator instructions
* Patient agrees to comply with the follow-up surveillance schedule
* Have ability to provide full written consent

Exclusion Criteria:

* High-risk cancer planned for neoadjuvant therapy
* Patients with a history of more than two weeks treatment with immunosuppressants (including systemic corticosteroids), cytotoxic chemotherapy within one month prior to initial screening, or who receive such medications during the screening period, or who are anticipated to require such medications during the course of the study
* Patients that have had prior hormonal therapy such as Lupron or oral antiandrogens ≤ 12 weeks prior to registration
* Clinical oligometastatic disease with > 3 nodes positive preoperative standard of care imaging of prostate region
* Previous history of pelvic radiation
* Patients with obesity defined as body mass index (BMI) > 40 kg/m^2
* History of prior laparoscopic inguinal hernia repair with mesh
* Scheduled at the time of screening to undergo chemotherapy, radiation, hormone therapy, or open surgery during the study period
* Inability to lie still for 75 minutes during 18F-rhPSMA-7.3 PSMA PET-MRI imaging
* Any neurologic disorder or psychiatric disorder that might confound postsurgical assessments
* Has any condition(s), which seriously compromises the subject's ability to participate in this study, sign consent, or has a known history of poor adherence with medical treatment
* Received administration of an investigational drug within 30 days prior to study registration, and/or has planned administration of another investigational product or procedure during participation in this study

Ages: 30 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-06-11 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of flotufolastat F-18 gallium (18F-rhPSMA-7.3) positron emission tomography (PET)/magnetic resonance (MRI) for the detection of lymph node metastasis | Up to 12 months
  Defined as the presence of lymph node positivity determined on final pathologic analysis compared to findings on preoperative 18F-rhPSMA-7.3 PSMA PET/MRI. Continuous variables will be summarized as mean (standard deviation) or median (range) while categorical variables will be reported as frequency (percentage).

SECONDARY OUTCOMES:
Specificity | Up to 12 months
  Defined as absence of lymph node metastasis on final pathologic analysis compared to findings on preoperative 18F-rhPSMA-7.3 PSMA PET/MRI.
Positive predictive value//negative predictive value (PPV/NPV) | Up to 120 months
  Defined as findings on 18F-rhPSMA-7.3 prostate specific membrane antigen (PSMA) PET/MRI compared to the presence or absence of lymph node metastasis on final pathologic analysis. Proportion of correct results will be compared between rhPSMA-7.3(18F) PET/MRI and the standard care.
Prostate specific antigen (PSA): < 5, 5-10, 10-20, > 20 | Up to 12 months
  Will investigate the impact of PSA as a clinicopathologic variable on lymph node metastasis when used alone and in combination with PSMA PET/MRI using 18F-rhPSMA-7.3.
Gleason score | Up to 12 months
  Will investigate the impact of Gleason score as a clinicopathologic variable on lymph node metastasis when used alone and in combination with PSMA PET/MRI using 18F-rhPSMA-7.3. Gleason score is a grading system for prostate cancer ranging from 6 (low-grade cancer) to 10 (high-grade cancer).
Digital rectal examination | Up to 12 months
  Will investigate the impact of digital rectal examination as clinicopathologic variable on lymph node metastasis when used alone and in combination with PSMA PET/MRI using 18F-rhPSMA-7.3.
Number of patients where management has changed | Up to 12 months
  Defined by the number of patients where PSMA PET/MRI depicts metastatic lesions (e.g. visceral/skeletal) or suspicious lymph nodes outside the true pelvis where standard of care imaging was negative. Proportion of correct results will be compared between rhPSMA-7.3(18F) PET/MRI and the standard care.
Rates of biochemical recurrent disease (BCR) | Up to 12 months
  BCR rates will be defined as PSA > 0.20 between patients with either negative or positive evidence of PSMA avid disease as indicated on the 18F-rhPSMA-7.3 PSMA PET /MRI and correlated to historical controls. Patients with positive and negative preop imaging results will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Ram A. Pathak, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials